CLINICAL TRIAL: NCT02891837
Title: A Phase III Double-Blind, Randomized, Placebo Controlled, Multi-Center Clinical Study to Evaluate the Efficacy and Safety of Intravenous L-citrulline for the Prevention of Clinical Sequelae of Acute Lung Injury Induced by Cardiopulmonary Bypass in Pediatric Subjects Undergoing Surgery for Congenital Heart Defects
Brief Title: L-citrulline for Prevention of Sequelae of Acute Lung Injury in Pediatrics Undergoing Cardiopulmonary Bypass for Heart Defects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asklepion Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CIT-003-01; 2016-002427-28 (EudraCT Number)
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Results first posted 2023-02-23 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-01

CONDITIONS: Acute Lung Injury
Keywords: L-citrulline; pediatric; Lung Injury; Bypass; Heart Defects; Clinical Sequelae
MeSH Terms: conditions — Acute Lung Injury; Lung Injury | interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-citrulline (Experimental): * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Interventions: Drug: L-citrulline
- Placebo (Placebo Comparator): * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: L-citrulline — * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Arms: L-citrulline
Other: Placebo — * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether L-citrulline is effective and safe in the prevention of clinical sequelae of Acute Lung Injury in pediatric subjects undergoing surgery for congenital heart defects.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo controlled, multicenter study that will compare the efficacy and safety of L-citrulline versus placebo in subjects undergoing surgery for congenital heart defects.

Eligible subjects undergoing repair of a large unrestrictive ventricular septal defect (VSD), a partial or complete atrioventricular septal defect (AVSD), or an ostium primum atrial septal defect (primum ASD) will be eligible for enrollment in this study.

Each enrolled subject will be randomized to receive either L-citrulline or placebo throughout all administrations in the study. Subjects will receive an L-citrulline bolus of 150 mg/kg or placebo at the initiation of cardiopulmonary bypass, the addition of L-citrulline at a concentration of 200 μmol/L or placebo given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L. L-citrulline bolus of 20 mg/kg or placebo 30 minutes after decannulation from cardiopulmonary bypass, followed immediately by a 9 mg/kg/hr continuous L-citrulline infusion or placebo for up to 48 hours.

The study drug or placebo infusion will be discontinued once invasive arterial blood pressure monitoring is discontinued or at 48 hours, whichever comes first. Subjects will be followed until Day 28 or discharge from the hospital, whichever comes first. For subjects discharged prior to Day 28, a final assessment via telephone will be conducted at Day 28.

ELIGIBILITY:
Inclusion Criteria:

* Subjects, parents, or legal guardian of the subject who are willing and able to sign informed consent
* Male and female subjects aged ≤18 years of age
* Infants, children and adolescents undergoing cardiopulmonary bypass (CPB) for repair of a large unrestrictive VSD, an ostium primum ASD, or a partial or complete AVSD
* Pre-operative echocardiogram which confirms the cardiovascular anatomy and defect to be surgically repaired

Exclusion Criteria:

* Evidence of pulmonary artery or vein abnormalities on the pre-operative echocardiogram that will not be addressed surgically. Specific abnormalities excluded include the following:

  * Significant pulmonary artery narrowing not amenable to surgical correction
  * Previous pulmonary artery stent placement
  * Significant left sided AV valve regurgitation not amenable to surgical correction
  * Pulmonary venous return abnormalities not amenable to surgical correction
  * Pulmonary vein stenosis not amenable to surgical correction
* Preoperative requirement for mechanical ventilation or intravenous inotrope support
* Presence of fixed or idiopathic pulmonary hypertension (i.e. Eisenmenger's Syndrome) prior to surgical repair
* Pre-operative use of medications to treat pulmonary hypertension
* Pregnancy; Females of child-bearing potential must be willing to participate an acceptable method of birth control for the duration of study participation (e.g. oral contraceptive, hormonal implant, intra-uterine device)
* Any condition which, in the opinion of the investigator, might interfere with the study objectives
* Participation in another clinical trial within 30 days of Screening or while participating in the current study, including the 28 days of follow-up post study drug administration

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 189 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gurdyal Kalsi, MD, Study Director — Asklepion Pharmaceuticals, LLC
Locations (29):
- United States (20):
  - University of Alabama, Birmingham, Alabama
  - Loma Linda University Children's Hospital, Loma Linda, California
  - University of California Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Nicklaus Children's Hospital, Miami, Florida
  - Arnold Palmer Hospital for Children, Orlando, Florida
  - Advocate Children's Hospital, Oak Lawn, Illinois
  - Riley Hospital for Children at Indiana University, Indianapolis, Indiana
  - The Johns Hopkins Hospital, Baltimore, Maryland
  - University of Mississippi Medical Center, Jackson, Mississippi
  - St Louis University, SSM Health Cardinal Glennon Children's Hospital, St Louis, Missouri
  - Washington University School of Medicine/ St Louis Children's Hospital, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - The Children's Hospital at Montefiore, The Bronx, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Primary Children's Hospital, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
- Austria (2):
  - LKH-Universitätsklinikum Graz Universitätsklinik für Kinder- und Jugendheilkunde, Graz
  - Medizinische Universität Wien, Klinik für Kinder- und Jugendheilkunde, Abteilung für Pädiatrische Kardiologie Kinderherzzentrum, Vienna
- Germany (4):
  - Universitätsmedizin Göttingen, Göttingen
  - Medizinische Hochschule Hannover, Hanover
  - Klinik für Kinderkardiologie und angeborene Herzfehler. Deutsches Herzzentrum München - Klinik an der TU München, München
  - Universitätsklinik Tübingen, Kinderkardiologie Pulmonologie, Intensivmedizin, Tübingen
- Israel (3):
  - Rambam Health Care Center, Haifa
  - Wolfson Medical Center, Holon
  - Sheba Medical Center, Ramat Gan

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- L-citrulline: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * L-citrulline at a concentration of 200 μmol/L given as a bolus during bypass. Administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
- Placebo: * Bolus at the initiation of cardiopulmonary bypass;
  * Bolus during bypass. Administered as a one-time bolus or multiple administrations during bypass;
  * Bolus 30 minutes after decannulation from cardiopulmonary bypass;
  * Continuous infusion for up to 48 hours.
Period: Overall Study
Arm/Group | L-citrulline | Placebo
Started | 99 | 90
Completed | 96 | 90
Not Completed | 3 | 0
Not completed — Lost to Follow-up | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Data shown for all patients (N=189). Additionally data are shown for patients within the USA only (N=137), a subset of all patients (N=189), because endpoints did not appear valid ex-US due to differences in standard of care.
  The estimated enrollment period was 11 months. The total trial period for a patient was up to 42 days (up to 2 weeks screening, 2 days treatment, up to 28 days follow-up). The trial end was defined as "last patient out" (LPO).
Groups:
- L-citrulline: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  L-citrulline: -Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
- Placebo: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Placebo: -Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
- Total: Total of all reporting groups
Arm/Group | L-citrulline | Placebo | Total
Number analyzed (Participants) | 99 | 90 | 189
Age, Customized [Mean (Standard Deviation); unit: Months] — Population: See section "Baseline Analysis Population Description".
  Months
    US Patients off mechanical ventilation in ≤48 hours: number analyzed (Participants) | 58 | 54 | 112
    US Patients off mechanical ventilation in ≤48 hours | 16.6 (28.4) | 17.3 (29.1) | 16.9 (28.6)
    US Patients off mechanical ventilation in >48 hours: number analyzed (Participants) | 13 | 12 | 25
    US Patients off mechanical ventilation in >48 hours | 6.6 (6.7) | 9.0 (11.9) | 7.8 (9.4)
    All patients | 17.4 (26.9) | 19.5 (31.6) | 18.4 (29.2)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: See section "Baseline Analysis Population Description".
  Participants
    USA patients: number analyzed (Participants) | 58 | 54 | 112
    USA patients: Female | 24 | 32 | 56
    USA patients: Male | 34 | 22 | 56
    All patients: Female | 45 | 53 | 98
    All patients: Male | 54 | 37 | 91
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: See section "Baseline Analysis Population Description".
  Participants
    USA patients: number analyzed (Participants) | 58 | 54 | 112
    USA patients: Hispanic or Latino | 5 | 8 | 13
    USA patients: Not Hispanic or Latino | 53 | 45 | 98
    USA patients: Unknown or Not Reported | 0 | 1 | 1
    All patients: Hispanic or Latino | 8 | 12 | 20
    All patients: Not Hispanic or Latino | 91 | 77 | 168
    All patients: Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 66 | 71 | 137
  Israel | 19 | 22 | 41
  Europe | 5 | 6 | 11

OUTCOME MEASURES:

1. Primary Outcome: A Composite Variable Consisting of the Longer of Either (1) Length of Time on Mechanical Ventilation or (2) Length of Inotrope Use.
Description: Mechanical ventilation (MV) = invasive or noninvasive MV incl. bilevel (biphasic) positive airway pressure or continuous positive airway pressure. Inotrope use = medications considered within the derivation of total inotrope score (dopamine, dobutamine, milrinone, epinephrine, phenylephrine, norepinephrine). Both measures recorded until earliest of subject hospital discharge or Day 28.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 3351.1 (5230.8) | 3549.6 (6069.1)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.4930, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Length of Time on Mechanical Ventilation
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 2398.4 (2031.8) | 5236.9 (4714.7)

3. Secondary Outcome: Length of Time on Positive Pressure Ventilation
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 2018.7 (4918.5) | 1285.6 (2354.8)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.1924, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Length of Time of Inotrope Use
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 2726.4 (3637.5) | 3167.3 (6035.2)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.8678, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Inotrope Score
Description: Inotrope score is reflective of the pharmacological support required by the cardiovascular system and is a good predictor of mortality and morbidity in patients undergoing bypass surgery. A lower inotrope score represents less pharmacological support and would indicate a lower risk for a poor clinical outcome. Therefore, any treatment effect would be indicated by a lower inotrope score in the citrulline group when compared to the placebo group.
  In this study, the score was calculated each hour post-operatively from the time of separation from bypass until the completion of study drug. Additionally, the total inotrope score over time until Day 28 or hospital discharge was derived. Inotrope score was calculated using the following formula:
  Total inotrope score = Dopamine dose (µg/kg/min) + Dobutamine dose (µg/kg/min) + 10 * Milrinone dose (µg/kg/min) + 100 * Epinephrine dose (µg/kg/min) + 100 * Phenylephrine dose (µg/kg/min) + 100 * Norepinephrine dose (µg/kg/min).
Time Frame: Up to 48 hours after separation from CBP
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: µg/kg/min
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
µg/kg/min
  1 hour after separation from CBP: number analyzed (Participants) | 99 | 86
  1 hour after separation from CBP | 1691.6 (11420.8) | 583.6 (4879.0)
  2 hours after separation from CBP: number analyzed (Participants) | 99 | 86
  2 hours after separation from CBP | 5076.2 (38880.0) | 537.1 (4870.3)
  3 hours after separation from CBP: number analyzed (Participants) | 99 | 88
  3 hours after separation from CBP | 5983.4 (39369.2) | 1258.2 (11744.0)
  4 hours after separation from CBP: number analyzed (Participants) | 98 | 88
  4 hours after separation from CBP | 6044.1 (39566.9) | 1257.4 (11744.1)
  5 hours after separation from CBP: number analyzed (Participants) | 98 | 88
  5 hours after separation from CBP | 6044.0 (39567.0) | 1257.3 (11744.1)
  6 hours after separation from CBP: number analyzed (Participants) | 99 | 89
  6 hours after separation from CBP | 5983.5 (39369.2) | 1243.4 (11677.9)
  7 hours after separation from CBP: number analyzed (Participants) | 99 | 89
  7 hours after separation from CBP | 5983.3 (39369.2) | 1243.4 (11677.9)
  8 hours after separation from CBP | 5983.2 (2007.7) | 39369.2 (13688.2)
  9 hours after separation from CBP | 5983.4 (39369.2) | 2007.1 (13688.3)
  10 hours after separation from CBP | 5983.0 (39369.3) | 2007.0 (13688.4)
  11 hours after separation from CBP | 5983.1 (39369.2) | 2007.0 (13688.4)
  12 hours after separation from CBP | 5983.5 (39369.2) | 2006.8 (13688.4)
  13 hours after separation from CBP | 5983.1 (39369.2) | 2006.7 (13688.4)
  14 hours after separation from CBP | 3255.8 (16449.2) | 2006.6 (13688.4)
  15 hours after separation from CBP | 3255.8 (16449.2) | 2006.5 (13688.4)
  16 hours after separation from CBP | 3255.4 (16449.2) | 2006.6 (13688.4)
  17 hours after separation from CBP | 3255.7 (16449.2) | 2006.5 (13688.4)
  18 hours after separation from CBP | 3255.4 (16449.2) | 2006.2 (13688.5)
  19 hours after separation from CBP | 3254.9 (16449.3) | 2006.1 (13688.5)
  20 hours after separation from CBP | 3254.9 (16449.3) | 2005.7 (13688.5)
  21 hours after separation from CBP | 2143.6 (12376.3) | 2107.8 (13707.6)
  22 hours after separation from CBP | 2143.2 (12376.3) | 2005.7 (13688.5)
  23 hours after separation from CBP | 2143.2 (12376.3) | 2005.6 (13688.6)
  24 hours after separation from CBP | 2143.0 (12376.4) | 2005.3 (13688.6)
  25 hours after separation from CBP | 2142.8 (12376.4) | 2005.2 (13688.6)
  26 hours after separation from CBP | 2142.8 (12376.4) | 2004.9 (13688.7)
  27 hours after separation from CBP | 2041.4 (2004.9) | 12352.5 (13688.7)
  28 hours after separation from CBP | 2041.1 (12352.5) | 2005.4 (13688.6)
  29 hours after separation from CBP | 2041.1 (12352.5) | 2004.7 (13688.7)
  30 hours after separation from CBP | 2041.1 (12352.5) | 2004.7 (13688.7)
  31 hours after separation from CBP | 2040.9 (12352.6) | 2004.6 (13688.7)
  32 hours after separation from CBP | 2041.0 (12352.5) | 2004.7 (13688.7)
  33 hours after separation from CBP | 2041.1 (12352.5) | 2004.6 (13688.7)
  34 hours after separation from CBP | 2041.0 (12352.5) | 2004.6 (13688.7)
  35 hours after separation from CBP | 2040.9 (12352.5) | 2004.4 (13688.7)
  36 hours after separation from CBP | 2041.1 (12352.5) | 2004.5 (13688.7)
  37 hours after separation from CBP | 2040.9 (12352.5) | 2004.4 (13688.7)
  38 hours after separation from CBP | 2040.9 (12352.6) | 2004.4 (13688.7)
  39 hours after separation from CBP | 2040.9 (12352.6) | 2004.3 (13688.7)
  40 hours after separation from CBP | 1012.5 (7071.8) | 2004.3 (13688.8)
  41 hours after separation from CBP | 1012.5 (7071.8) | 1282.1 (8736.4)
  42 hours after separation from CBP | 1012.5 (7071.8) | 780.0 (7378.4)
  43 hours after separation from CBP | 1012.4 (7071.8) | 779.9 (7378.4)
  44 hours after separation from CBP | 1012.4 (7071.8) | 780.1 (7378.4)
  45 hours after separation from CBP | 1012.3 (7071.8) | 780.0 (7378.4)
  46 hours after separation from CBP | 1012.1 (7071.9) | 780.0 (7378.4)
  47 hours after separation from CBP | 1012.1 (7071.8) | 780.0 (7378.4)
  48 hours after separation from CBP | 1012.1 (7071.9) | 779.8 (7378.4)

6. Secondary Outcome: Hemodynamic Improvement: Heart Rate
Description: Heart rate at hours 1, 2, 4, 12, 24 and 48.
Time Frame: 2 Days
Population: Modified FAS
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Beats per minute
  1 hour: number analyzed (Participants) | 96 | 88
  1 hour | 80.1 (67.9) | 83.6 (60.1)
  2 hours: number analyzed (Participants) | 95 | 87
  2 hours | 111.2 (45.7) | 116.0 (46.7)
  4 hours: number analyzed (Participants) | 96 | 86
  4 hours | 130.4 (27.7) | 133.5 (20.1)
  12 hours | 120.9 (22.0) | 161.9 (17.6)
  24 hours: number analyzed (Participants) | 99 | 89
  24 hours | 122.2 (22.2) | 118.3 (14.9)
  48 hours: number analyzed (Participants) | 93 | 79
  48 hours | 125.9 (18.7) | 125.4 (21.0)

7. Secondary Outcome: Hemodynamic Improvement: Systemic Arterial Blood Pressure
Description: Systemic arterial blood pressure at hours 1, 2, 4, 12, 24 and 48.
Time Frame: 2 Days
Population: Modified FAS
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Millimeters of mercury
  1 hour: number analyzed (Participants) | 94 | 86
  1 hour | 18.4 (16.2) | 15.3 (14.9)
  2 hours: number analyzed (Participants) | 94 | 85
  2 hours | 31.7 (17.9) | 32.5 (18.2)
  4 hours: number analyzed (Participants) | 95 | 85
  4 hours | 42.4 (12.1) | 42.1 (12.3)
  12 hours: number analyzed (Participants) | 94 | 89
  12 hours | 39.7 (12.1) | 40.7 (10.6)
  24 hours: number analyzed (Participants) | 90 | 86
  24 hours | 41.0 (12.2) | 40.1 (10.8)
  48 hours: number analyzed (Participants) | 54 | 45
  48 hours | 40.3 (15.8) | 42.1 (11.6)

8. Secondary Outcome: Hemodynamic Improvement: Oxygen Saturation
Description: Oxygen saturation at hours 1, 2, 4, 12, 24 and 48.
Time Frame: 2 Days
Population: Modified FAS
Measure: Mean (Standard Deviation); unit: Percentage of hemoglobin bound to oxygen
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Percentage of hemoglobin bound to oxygen
  1 hour: number analyzed (Participants) | 95 | 89
  1 hour | 97.2 (7.9) | 95.7 (15.8)
  2 hours: number analyzed (Participants) | 95 | 90
  2 hours | 98.6 (4.6) | 97.6 (10.7)
  4 hours: number analyzed (Participants) | 95 | 86
  4 hours | 98.5 (2.1) | 98.1 (2.7)
  12 hours: number analyzed (Participants) | 98 | 90
  12 hours | 97.9 (2.4) | 97.6 (2.6)
  24 hours: number analyzed (Participants) | 99 | 88
  24 hours | 97.1 (4.0) | 97.6 (2.7)
  48 hours: number analyzed (Participants) | 95 | 79
  48 hours | 97.6 (2.8) | 97.8 (2.6)

9. Secondary Outcome: Hemodynamic Improvement: Central Venous Pressure
Description: Central venous pressure at hours 1, 2, 4, 12, 24 and 48.
Time Frame: 2 Days
Population: Modified FAS
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Millimeters of mercury
  1 hour: number analyzed (Participants) | 69 | 61
  1 hour | 10.2 (20.1) | 12.9 (28.0)
  72 hours: number analyzed (Participants) | 79 | 72
  72 hours | 10.3 (5.6) | 13.2 (23.9)
  4 hours: number analyzed (Participants) | 81 | 75
  4 hours | 13.1 (23.7) | 13.2 (27.4)
  12 hours: number analyzed (Participants) | 72 | 69
  12 hours | 9.7 (4.1) | 9.0 (3.6)
  24 hours: number analyzed (Participants) | 64 | 64
  24 hours | 10.9 (5.4) | 9.8 (3.6)
  48 hours: number analyzed (Participants) | 35 | 28
  48 hours | 11.8 (6.2) | 9.6 (8.3)

10. Secondary Outcome: Thoracotomy Output
Description: The thoracotomy output is defined as the total volume of chest tube drainage recorded in cc prior to discontinuation of chest intubation. The total postoperative duration (in hours) that the chest tube is used will be calculated as the time from the end of the surgery to the time the chest tube is removed. If an additional chest tube is required or reinserted (until discharge from the hospital or at Day 28) the duration that the additional chest tube was used (from time of insertion to time of removal) will be added to the time the original chest tube was used for the total postoperative duration. If a subject did not use any chest tube the duration is set to 0. As a sensitivity analysis, subjects with no use of chest tube will be excluded. For subjects who died before discharge from the hospital or before Day 28, respectively, the observed duration of chest tube drainage will be used.
Time Frame: 28 Days
Population: Modified FAS
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Milliliters | 206.41 (137.26) | 198.94 (143.85)

11. Secondary Outcome: Length of Time of Intubation
Description: The length will be derived as the time in hours from separation from CPB until discontinuation of intubation. Any duration of re-use of intubation will continue to accrue. If a subject did not use any intubation the length is set to 0. As a sensitivity analysis, subjects with no use of intubations will be excluded. For subjects who died before discharge from the hospital or before Day 28, respectively, the observed length of time on intubation will be used. As sensitivity analyses subjects who died will (1) be excluded from analysis and (2) be assigned a length of time on intubation of 28 days.
  For the length of time on intubation the same analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 1600.4 (4488.9) | 1303.9 (4408.3)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.6422, Wilcoxon (Mann-Whitney)

12. Secondary Outcome: Length of Pediatric Intensive Care Unit (PICU) Stay
Description: The length of PICU stay will be calculated as the total number of days postoperative until discharge from PICU. For subjects who died before discharge from PICU or before Day 28, respectively, the observed length of PICU stay will be used. As sensitivity analyses subjects who died will (1) be excluded from analysis and (2) be assigned a length of PICU stay of 28 days. For the length of PICU stay the same analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Days | 6.3 (8.5) | 6.5 (9.2)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.7572, Wilcoxon (Mann-Whitney)

13. Secondary Outcome: Length of Time on Vasodilators
Description: Length of time on vasodilators will be measured from first use following separation from bypass, until the subject is discharged from the hospital or at Day 28. The length will be derived as the time in hours from separation from CPB until discontinuation of all vasodilators.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Minutes | 1668.4 (5751.6) | 611.3 (1212.5)

14. Secondary Outcome: Length of Hospitalization
Description: The length of hospitalization will be calculated as the total number of days postoperative until discharge from the hospital. For subjects who died before discharge from the hospital or before Day 28, respectively, the observed length of hospitalization will be used. As sensitivity analyses subjects who died will (1) be excluded from analysis and (2) be assigned a length of hospitalization of 28 days. The same analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Days | 7.1 (5.1) | 3.9 (3.9)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Test type: Other; p = 0.3681, Wilcoxon (Mann-Whitney)

15. Secondary Outcome: Patients With Plasma Concentrations of Citrulline
Description: Plasma citrulline concentrations will be assessed in both treatment groups to determine the number of patients who reach the therapeutic sustained target plasma citrulline level of ≥100 μmol/L. Blood collection for assessment of plasma citrulline concentrations will be taken prior to surgery, during surgery, 30 minutes post-decannulation after CPB (prior to bolus and 5 minutes after bolus), at the specified post-operative time points (6h, 12h, 24h, 48h), and at hospital discharge or Day 28, whichever occurs first.
Time Frame: 28 Days
Population: All patients (mFAS)
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
umol/L
  Day 0 - Intra-Op: number analyzed (Participants) | 99 | 89
  Day 0 - Intra-Op | 2179.6 (1046.8) | 26.4 (9.1)
  Day 0 - 0 hours (prior to bolus): number analyzed (Participants) | 99 | 88
  Day 0 - 0 hours (prior to bolus) | 1808.9 (12549.4) | 27.6 (11.3)
  Day 0 - 0 hours (post bolus): number analyzed (Participants) | 98 | 89
  Day 0 - 0 hours (post bolus) | 1387.8 (4957.5) | 27.8 (11.6)
  Day 0 - 6 hours: number analyzed (Participants) | 98 | 87
  Day 0 - 6 hours | 146.6 (67.3) | 20.3 (10.2)
  Day 0 - 12 hours: number analyzed (Participants) | 96 | 87
  Day 0 - 12 hours | 123.8 (41.3) | 18.5 (8.4)
  Day 1 - 24 hours: number analyzed (Participants) | 92 | 84
  Day 1 - 24 hours | 102.1 (42.6) | 14.9 (6.8)
  Day 2 - 48 hours: number analyzed (Participants) | 53 | 51
  Day 2 - 48 hours | 68.2 (44.9) | 12.1 (5.8)
  Day 28/ Discharge: number analyzed (Participants) | 26 | 24
  Day 28/ Discharge | 21.9 (29.5) | 16.9 (6.2)

16. Secondary Outcome: Occurrence of Adverse and Serious Adverse Events
Description: Pre-treatment adverse events and treatment adverse events will be analyzed separately. The number of affected subjects will be reported.
Time Frame: 28 Days
Population: The analysis of AEs included all patients who were randomized, underwent surgery and received study medication
Measure: Count of Participants; unit: Participants
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Participants
  Any adverse event | 68 | 62
  Pre-treatment adverse events | 19 | 12
  Treatment emergent adverse events | 68 | 61
  Any serious adverse event | 11 | 6

17. Secondary Outcome: Number of Patients With Refractory Hypotension
Description: Refractory hypotension is defined as a 20% drop of mean arterial pressure (MAP) below specific age-related criteria for more than 30 minutes. The number of subjects with any refractory hypotension from end of surgery until 48 hours will be compared between groups.
Time Frame: 2 Days
Population: SAF
Measure: Count of Participants; unit: Participants
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 99 | 90
Participants | 0 | 0

18. Post Hoc Outcome: A Composite Variable Consisting of the Longer of Either (1) Length of Time on Mechanical Ventilation or (2) Length of Inotrope Use.
Description: Mechanical ventilation (MV) = invasive or noninvasive MV incl. bilevel (biphasic) positive airway pressure or continuous positive airway pressure. Inotrope use = medications considered within the derivation of total inotrope score (dopamine, dobutamine, milrinone, epinephrine, phenylephrine, norepinephrine). Both measures recorded until earliest of subject hospital discharge or Day 28.
  Note: data are reported for post-hoc analyses based on a modified full analysis set (mFAS) targeting the US population for a 48-hour treatment period. Analysis method used was quartiles based, but followed prescribed statistical analysis plan methods. This is because chosen endpoints did not appear to be valid in the ex-US population due to differences in physician decision making. In the US, extubation occurs as soon as a patient's physical condition permits (only more severely ill children remain on mechanical ventilation); conversely, in ex-US sites, children remain on mechanical ventilation.
Time Frame: 28 Days
Population: Only data from US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 1484.9 (1317.1) | 1730.7 (1435.5)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; H0: Composite endpoint in L-citrulline group = placebo group H1: Composite endpoint in L-citrulline group ≠ placebo group H0 tested using Wilcoxon-rank-sum test. Significance level = 1% (2-sided); Test type: Other — Sample size calculated with nQuery 7.0. Assumed standard deviation = 50 h, & mean values of 44 h (placebo) & 14 h (L-citrulline group), estimated effect size = 0.600, yielding a sample size N=92/group (two-sided Wilcoxon-rank-sum test with 0.01 significance level and 90% power). Assumptions for standard deviation & mean based on Study CIT-002-01 results. To allow for subjects being enrolled but not assigned to the full analysis set (FAS), an overall N=95 subjects per group were to be enrolled; p = 0.1560, Wilcoxon (Mann-Whitney) — The threshold for statistical significance was p = 0.05; Location shift = 219.0, 95% CI 2-sided [-88.0 to 626.0] — Treatment difference = L-citrulline - placebo For the mean and median values, that the estimated values are given in minutes [min]
Statistical Analysis 2: Comparison: L-citrulline vs Placebo; Post hoc analyses were done for US patients on mechanical ventilation for <=48 hours. For all post hoc analyses a significance level of 5% was applied; Test type: Other; p = 0.1627, t-test, 2 sided — The threshold for statistical significance was 0.05; The results of the T-test should be interpreted with caution since the endpoint is not normally distributed; Location shift = 813.1, 95% CI 2-sided [-335.5 to 1961.6] — Treatment difference = L-citrulline - placebo. For the mean and median values, the estimated values are given in minutes

19. Post Hoc Outcome: Length of Time on Mechanical Ventilation
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 420.2 (585.1) | 649.7 (786.4)

20. Post Hoc Outcome: Length of Time on Positive Pressure Ventilation
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 200.9 (560.5) | 358.0 (758.5)

21. Post Hoc Outcome: Length of Time of Inotrope Use
Description: The same definitions and analyses as described for the primary endpoint will be applied.
Time Frame: 28 days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 1428.6 (1344.6) | 1653.1 (1485.7)

22. Post Hoc Outcome: Inotrope Score
Description: as for outcome 5
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: µg/kg/min
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
µg/kg/min
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after separation from CBP | 14.7 (43.0) | 17.4 (44.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after separation from CBP | 17.2 (98.0) | 13.5 (58.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 3 hours after separation from CBP | 4.5 (4.2) | 4.5 (3.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after separation from CBP | 3.6 (2.6) | 4.4 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 5 hours after separation from CBP | 3.7 (2.8) | 4.4 (2.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 6 hours after separation from CBP | 3.7 (2.8) | 4.4 (2.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 7 hours after separation from CBP | 3.6 (2.7) | 4.5 (3.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 8 hours after separation from CBP | 3.4 (2.4) | 4.5 (3.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 9 hours after separation from CBP | 3.4 (2.4) | 4.4 (3.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 10 hours after separation from CBP | 3.4 (2.4) | 4.3 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 11 hours after separation from CBP | 3.3 (2.5) | 4.1 (2.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after separation from CBP | 3.4 (3.5) | 4.0 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 13 hours after separation from CBP | 3.3 (2.8) | 3.8 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 14 hours after separation from CBP | 3.1 (2.5) | 3.7 (3.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 15 hours after separation from CBP | 3.1 (2.6) | 3.7 (3.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 16 hours after separation from CBP | 3.0 (2.6) | 3.5 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 17 hours after separation from CBP | 3.1 (2.8) | 3.8 (4.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 18 hours after separation from CBP | 3.0 (2.7) | 3.4 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 19 hours after separation from CBP | 2.8 (2.7) | 3.4 (3.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 20 hours after separation from CBP | 2.9 (3.2) | 3.1 (3.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 21 hours after separation from CBP | 2.6 (2.8) | 3.1 (3.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 22 hours after separation from CBP | 2.3 (2.7) | 2.7 (3.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 23 hours after separation from CBP | 2.2 (3.2) | 2.9 (4.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after separation from CBP | 2.1 (3.1) | 2.3 (3.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 25 hours after separation from CBP | 1.8 (2.6) | 2.4 (4.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 26 hours after separation from CBP | 1.7 (2.8) | 1.9 (3.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 27 hours after separation from CBP | 1.5 (2.7) | 1.8 (2.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 28 hours after separation from CBP | 1.4 (2.3) | 2.0 (3.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 29 hours after separation from CBP | 1.3 (2.3) | 1.5 (2.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 30 hours after separation from CBP | 1.4 (2.5) | 1.4 (2.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 31 hours after separation from CBP | 1.2 (2.3) | 1.4 (2.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 32 hours after separation from CBP | 1.2 (2.3) | 1.5 (3.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 33 hours after separation from CBP | 1.2 (2.4) | 1.4 (2.7)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 34 hours after separation from CBP | 1.1 (2.2) | 1.3 (2.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 35 hours after separation from CBP | 1.2 (2.3) | 1.2 (2.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 36 hours after separation from CBP | 1.1 (2.2) | 1.3 (2.7)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 37 hours after separation from CBP | 1.1 (2.3) | 1.2 (2.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 38 hours after separation from CBP | 1.0 (2.1) | 1.2 (2.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 39 hours after separation from CBP | 1.0 (2.1) | 1.1 (2.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 40 hours after separation from CBP | 1.0 (2.1) | 1.1 (2.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 41 hours after separation from CBP | 0.9 (2.1) | 1.1 (2.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 42 hours after separation from CBP | 1.0 (2.3) | 1.1 (2.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 43 hours after separation from CBP | 0.8 (1.9) | 1.0 (2.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 44 hours after separation from CBP | 0.9 (2.2) | 1.2 (2.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 45 hours after separation from CBP | 0.7 (2.0) | 1.0 (2.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 46 hours after separation from CBP | 0.6 (1.4) | 1.1 (2.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 47 hours after separation from CBP | 0.6 (1.4) | 1.0 (2.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after separation from CBP | 0.4 (1.2) | 0.7 (1.5)

23. Post Hoc Outcome: Hemodynamic Improvement: Heart Rate
Description: Heart rate will be calculated using the absolute changes from baseline at hours 1, 2, 4, 12, 24 and 48 and will be compared between groups using an ANOVA with a fixed effect for treatment group and baseline level. Summary tables describing descriptive measurements will be generated for absolute values and absolute change from baseline values for all observed time points.
Time Frame: 2 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 51 | 49
Beats per minute
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after surgery start | -43.9 (78.6) | -40.6 (66.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start: number analyzed (Participants) | 50 | 48
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start | -14.1 (50.0) | 1.1 (43.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start: number analyzed (Participants) | 48 | 48
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start | 10.0 (27.3) | 18.5 (24.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after surgery start | 1.8 (19.6) | 5.4 (16.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start: number analyzed (Participants) | 51 | 48
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start | 3.1 (21.3) | 3.3 (20.3)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start: number analyzed (Participants) | 46 | 40
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start | 5.8 (21.2) | 7.1 (26.6)

24. Post Hoc Outcome: Hemodynamic Improvement: Systemic Arterial Blood Pressure
Description: Systemic arterial blood pressure will be calculated using the absolute changes from baseline at hours 1, 2, 4, 12, 24 and 48 and will be compared between groups using an ANOVA with a fixed effect for treatment group and baseline level. Summary tables describing descriptive measurements will be generated for absolute values and absolute change from baseline values for all observed time points.
Time Frame: 2 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 49 | 48
Millimeters of mercury
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after surgery start | -17.9 (13.2) | -22.3 (17.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start: number analyzed (Participants) | 48 | 46
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start | -3.8 (19.1) | -4.0 (17.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start: number analyzed (Participants) | 48 | 47
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start | 7.3 (12.5) | 8.9 (13.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after surgery start | 6.6 (11.7) | 7.2 (13.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start: number analyzed (Participants) | 46 | 45
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start | 8.8 (12.9) | 8.4 (11.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start: number analyzed (Participants) | 21 | 19
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start | 6.5 (17.9) | 7.6 (14.5)

25. Post Hoc Outcome: Hemodynamic Improvement: Oxygen Saturation
Description: Oxygen saturation will be calculated using the absolute changes from baseline at hours 1, 2, 4, 12, 24 and 48 and will be compared between groups using an ANOVA with a fixed effect for treatment group and baseline level. Summary tables describing descriptive measurements will be generated for absolute values and absolute change from baseline values for all observed time points.
Time Frame: 2 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Percentage of hemoglobin bound to oxygen
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 51 | 49
Percentage of hemoglobin bound to oxygen
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after surgery start | 1.3 (6.2) | -1.8 (18.2)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start: number analyzed (Participants) | 49 | 49
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after surgery start | 2.3 (9.4) | 1.5 (9.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start: number analyzed (Participants) | 47 | 48
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after surgery start | 1.4 (8.8) | 0.7 (9.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after surgery start: number analyzed (Participants) | 50 | 49
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after surgery start | 0.8 (8.4) | 0.7 (8.7)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start: number analyzed (Participants) | 50 | 49
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after surgery start | -0.2 (9.9) | 0.2 (8.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start: number analyzed (Participants) | 48 | 40
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after surgery start | 0.4 (9.6) | 1.1 (10.3)

26. Post Hoc Outcome: Hemodynamic Improvement: Central Venous Pressure
Description: Central venous pressure will be calculated using the absolute changes from baseline at hours 1, 2, 4, 12, 24 and 48 and will be compared between groups using an ANOVA with a fixed effect for treatment group and baseline level. Summary tables describing descriptive measurements will be generated for absolute values and absolute change from baseline values for all observed time points.
Time Frame: 2 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 34 | 32
Millimeters of mercury
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after treatment: number analyzed (Participants) | 33 | 32
  Patients on mechanical ventilation for ≤48 hours (US patients) - 1 hour after treatment | -10.0 (48.8) | -6.8 (45.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after treatment: number analyzed (Participants) | 34 | 31
  Patients on mechanical ventilation for ≤48 hours (US patients) - 2 hours after treatment | -6.5 (47.4) | -5.2 (43.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after treatment: number analyzed (Participants) | 31 | 31
  Patients on mechanical ventilation for ≤48 hours (US patients) - 4 hours after treatment | 6.7 (36.5) | -5.2 (41.7)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after treatment: number analyzed (Participants) | 24 | 24
  Patients on mechanical ventilation for ≤48 hours (US patients) - 12 hours after treatment | -10.4 (58.6) | -7.7 (41.1)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after treatment: number analyzed (Participants) | 19 | 22
  Patients on mechanical ventilation for ≤48 hours (US patients) - 24 hours after treatment | -0.1 (11.2) | -8.3 (43.9)
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after treatment: number analyzed (Participants) | 6 | 5
  Patients on mechanical ventilation for ≤48 hours (US patients) - 48 hours after treatment | -5.3 (17.3) | 6.2 (20.8)
Statistical Analysis 1: Comparison: L-citrulline vs Placebo; Values at 48 hours post-surgery start for all US patients on ventilation for ≤48 hours are presented. Treatment group, baseline values and site were included as fixed factors, site*treatment as interaction terms in this ANOVA. The normality assumption of residuals is critical for all considered timepoints. Please interpret results with caution; Test type: Other; p = 0.0326, ANOVA — The threshold for statistical significance was 0.05
Statistical Analysis 2: Comparison: L-citrulline vs Placebo; Values at 48 hours post-surgery start for ALL patients on ventilation for ≤48 hours are presented. Treatment group, baseline values and site were included as fixed factors, site*treatment as interaction terms in this ANOVA. The normality assumption of residuals is critical for all considered timepoints. Please interpret results with caution; Test type: Other; p = 0.0026, ANOVA — The threshold for statistical significance was 0.05

27. Post Hoc Outcome: Thoracotomy Output
Description: as for outcome 10
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Milliliters
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Milliliters | 209.42 (141.35) | 194.35 (124.41)

28. Post Hoc Outcome: Length of Time of Intubation
Description: as for outcome 11
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 329.9 (432.6) | 386.5 (556.6)

29. Post Hoc Outcome: Length of Pediatric Intensive Care Unit (PICU) Stay
Description: as for outcome 12
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 51 | 50
Days | 5.6 (9.2) | 7.1 (10.7)

30. Post Hoc Outcome: Length of Time on Vasodilators
Description: as for outcome 13
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Minutes | 617.9 (910.0) | 624.8 (1077.1)

31. Post Hoc Outcome: Length of Hospitalization
Description: as for outcome 14
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
Days | 4.9 (2.6) | 4.8 (2.5)

32. Post Hoc Outcome: Patients With Plasma Concentrations of Citrulline
Description: as for outcome 15
Time Frame: 28 Days
Population: Only US patients on mechanical ventilation for ≤48 hours are analysed.
Measure: Mean (Standard Deviation); unit: umol/L
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 58 | 54
umol/L
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - Intra-Op | 2264.6 (890.1) | 26.7 (9.5)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 0 hours (prior to bolus): number analyzed (Participants) | 58 | 53
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 0 hours (prior to bolus) | 2625.4 (16391.9) | 25.4 (8.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 0 hours (post bolus): number analyzed (Participants) | 57 | 54
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 0 hours (post bolus) | 760.1 (369.5) | 25.7 (9.0)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 6 hours | 133.7 (39.2) | 18.8 (8.6)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 12 hours: number analyzed (Participants) | 57 | 54
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 0 - 12 hours | 125.6 (32.9) | 17.6 (7.4)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 1 - 24 hours: number analyzed (Participants) | 54 | 50
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 1 - 24 hours | 108.4 (43.0) | 14.6 (6.6)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 2 - 48 hours: number analyzed (Participants) | 23 | 21
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 2 - 48 hours | 73.3 (49.6) | 12.4 (6.8)
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 28/ Discharge: number analyzed (Participants) | 11 | 9
  Patients on mechanical ventilation for ≤48 hours (US patients) - Day 28/ Discharge | 28.5 (44.3) | 16.2 (6.4)

33. Post Hoc Outcome: Occurrence of Adverse and Serious Adverse Events
Description: Pre-treatment adverse events and treatment adverse events will be analyzed separately. The number affected subjects will be reported.
Time Frame: 28 Days
Population: The analysis of AEs included all patients who were randomized, underwent surgery and received study medication divided into the following subgroups:
  * All patients off mechanical ventilation in ≤48 hours (N=147)
  * US patients off mechanical ventilation in ≤48 hours (N=112)
  * All patients off mechanical ventilation in >48 hours (N=42)
  * US patients off mechanical ventilation in >48 hours (N=25)
Measure: Count of Participants; unit: Participants
Groups:
- L-citrulline - All Patients Off Mechanical Ventilation in ≤48 Hours; L-citrulline - US Patients Off Mechanical Ventilation in ≤48 Hours; L-citrulline - All Patients Off Mechanical Ventilation in >48 Hours; L-citrulline - US Patients Off Mechanical Ventilation in >48 Hours: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * L-citrulline at a concentration of 200 μmol/L given as a bolus during bypass. Administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
- Placebo - All Patients Off Mechanical Ventilation in ≤48 Hours; Placebo - US Patients Off Mechanical Ventilation in ≤48 Hours; Placebo - All Patients Off Mechanical Ventilation in >48 Hours; Placebo - US Patients Off Mechanical Ventilation in >48 Hours: * Bolus at the initiation of cardiopulmonary bypass;
  * Bolus during bypass. Administered as a one-time bolus or multiple administrations during bypass;
  * Bolus 30 minutes after decannulation from cardiopulmonary bypass;
  * Continuous infusion for up to 48 hours.
Arm/Group | L-citrulline - All Patients Off Mechanical Ventilation in ≤48 Hours | L-citrulline - US Patients Off Mechanical Ventilation in ≤48 Hours | L-citrulline - All Patients Off Mechanical Ventilation in >48 Hours | L-citrulline - US Patients Off Mechanical Ventilation in >48 Hours | Placebo - All Patients Off Mechanical Ventilation in ≤48 Hours | Placebo - US Patients Off Mechanical Ventilation in ≤48 Hours | Placebo - All Patients Off Mechanical Ventilation in >48 Hours | Placebo - US Patients Off Mechanical Ventilation in >48 Hours
Number analyzed (Participants) | 76 | 58 | 23 | 13 | 71 | 54 | 19 | 12
Participants
  Any adverse event | 48 | 30 | 20 | 10 | 47 | 30 | 15 | 8
  Pre-treatment adverse events | 12 | 6 | 7 | 3 | 9 | 6 | 3 | 1
  Treatment emergent adverse events | 48 | 30 | 20 | 10 | 46 | 29 | 15 | 8
  Any serious adverse event | 4 | 2 | 7 | 4 | 2 | 2 | 4 | 3
  Pre-treatment serious adverse events | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 0
  Treatment-emergent serious adverse events | 4 | 2 | 7 | 4 | 2 | 2 | 4 | 3

34. Post Hoc Outcome: Number of Patients With Refractory Hypotension
Description: as for outcome 17
Time Frame: 2 Days
Population: Data not available for this endpoint. Full analysis to include all secondary endpoints was not feasible and not done. Several post-hoc analysis were instead conducted on the primary endpoint and presented to the FDA.
Arm/Group | L-citrulline | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the time of giving informed consent until the Day 28 telephone follow-up.
Groups:
- L-citrulline - All Patients; L-citrulline - All Patients on Mechanical Ventilation for ≤48 Hours; L-citrulline - US Patients on Mechanical Ventilation for ≤48 Hours; L-citrulline - All Patients on Mechanical Ventilation for >48 Hours; L-citrulline - US Patients on Mechanical Ventilation for >48 Hours: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  L-citrulline: -Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass, but after removal of any crystalloid base;
  * Addition of study medication at a concentration of 200 μmol/L given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations to compensate for fluids containing L-citrulline that may be removed from the patient during the course of the operation and thus to maintain the concentration of 200 μmol/L;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
- Placebo - All Patients; Placebo - All Patients on Mechanical Ventilation for ≤48 Hours; Placebo - US Patients on Mechanical Ventilation for ≤48 Hours; Placebo - All Patients on Mechanical Ventilation for >48 Hours; Placebo - US Patients on Mechanical Ventilation for >48 Hours: * Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
  Placebo: -Bolus of 150 mg/kg at the initiation of cardiopulmonary bypass;
  * Addition of placebo matched for volume given as a bolus during bypass. This may be administered as a one-time bolus or multiple administrations during bypass;
  * Bolus of 20 mg/kg 30 minutes after decannulation from cardiopulmonary bypass;
  * 9 mg/kg/hr continuous infusion for up to 48 hours.
Arm/Group | L-citrulline - All Patients | Placebo - All Patients | L-citrulline - All Patients on Mechanical Ventilation for ≤48 Hours | L-citrulline - US Patients on Mechanical Ventilation for ≤48 Hours | L-citrulline - All Patients on Mechanical Ventilation for >48 Hours | L-citrulline - US Patients on Mechanical Ventilation for >48 Hours | Placebo - All Patients on Mechanical Ventilation for ≤48 Hours | Placebo - US Patients on Mechanical Ventilation for ≤48 Hours | Placebo - All Patients on Mechanical Ventilation for >48 Hours | Placebo - US Patients on Mechanical Ventilation for >48 Hours
All-Cause Mortality (participants affected / at risk) | 0/99 | 0/90 | 0/76 | 0/58 | 0/23 | 0/13 | 0/71 | 0/54 | 1/19 | 0/12
Serious Adverse Events (participants affected / at risk) | 11/99 | 6/90 | 5/76 | 2/58 | 7/23 | 4/13 | 2/71 | 2/54 | 4/19 | 3/12
Other Adverse Events (participants affected / at risk) | 68/99 | 61/90 | 48/76 | 30/58 | 20/23 | 10/13 | 46/71 | 29/54 | 15/19 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-citrulline - All Patients (N=99) | Placebo - All Patients (N=90) | L-citrulline - All Patients on Mechanical Ventilation for ≤48 Hours (N=76) | L-citrulline - US Patients on Mechanical Ventilation for ≤48 Hours (N=58) | L-citrulline - All Patients on Mechanical Ventilation for >48 Hours (N=23) | L-citrulline - US Patients on Mechanical Ventilation for >48 Hours (N=13) | Placebo - All Patients on Mechanical Ventilation for ≤48 Hours (N=71) | Placebo - US Patients on Mechanical Ventilation for ≤48 Hours (N=54) | Placebo - All Patients on Mechanical Ventilation for >48 Hours (N=19) | Placebo - US Patients on Mechanical Ventilation for >48 Hours (N=12)
Staphylococcal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac tamponade (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular fibrillation (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Feeding disorder (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Junctional ectopic tachycardia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Swallow study abnormal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | L-citrulline - All Patients (N=99) | Placebo - All Patients (N=90) | L-citrulline - All Patients on Mechanical Ventilation for ≤48 Hours (N=76) | L-citrulline - US Patients on Mechanical Ventilation for ≤48 Hours (N=58) | L-citrulline - All Patients on Mechanical Ventilation for >48 Hours (N=23) | L-citrulline - US Patients on Mechanical Ventilation for >48 Hours (N=13) | Placebo - All Patients on Mechanical Ventilation for ≤48 Hours (N=71) | Placebo - US Patients on Mechanical Ventilation for ≤48 Hours (N=54) | Placebo - All Patients on Mechanical Ventilation for >48 Hours (N=19) | Placebo - US Patients on Mechanical Ventilation for >48 Hours (N=12)
Tachycardia (Cardiac disorders) | 12 (12) | 4 (4) | 9 (9) | 3 (3) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 11 (11) | 16 (16) | 8 (8) | 4 (4) | 3 (3) | 0 (0) | 12 (12) | 7 (7) | 4 (4) | 2 (2)
Vomiting (Gastrointestinal disorders) | 6 (6) | 12 (13) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 10 (11) | 4 (4) | 2 (2) | 2 (2)
Pain (General disorders) | 16 (20) | 19 (34) | 11 (15) | 1 (1) | 5 (5) | 1 (1) | 16 (31) | 2 (3) | 3 (3) | 0 (0)
Pyrexia (General disorders) | 19 (28) | 13 (13) | 14 (22) | 2 (2) | 5 (6) | 2 (2) | 11 (11) | 3 (3) | 2 (2) | 1 (1)
Haemoglobin decreased (Investigations) | 7 (9) | 12 (12) | 6 (7) | 3 (3) | 1 (2) | 0 (0) | 10 (10) | 2 (2) | 2 (2) | 1 (1)
Electrolyte imbalance (Metabolism and nutrition disorders) | 6 (8) | 6 (7) | 4 (6) | 0 (0) | 2 (2) | 0 (0) | 5 (5) | 0 (0) | 1 (2) | 0 (0)
Hypocalcaemia (Investigations) | 7 (7) | 6 (6) | 5 (5) | 5 (5) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 3 (3) | 2 (2)
Hypokalaemia (Investigations) | 12 (12) | 15 (16) | 9 (9) | 5 (5) | 1 (1) | 2 (2) | 11 (11) | 9 (9) | 1 (1) | 1 (1)
Restlessness (Psychiatric disorders) | 14 (15) | 14 (14) | 8 (9) | 0 (0) | 6 (6) | 0 (0) | 10 (10) | 0 (0) | 4 (4) | 0 (0)
Metabolic acidosis (Metabolism and nutrition disorders) | 4 (4) | 6 (6) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 5 (5) | 0 (0) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 2 (2) | 4 (5) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 12 (13) | 11 (15) | 6 (6) | 1 (1) | 6 (7) | 2 (3) | 7 (8) | 2 (2) | 4 (7) | 0 (0)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 5 (6) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 6 (7) | 3 (3) | 0 (0) | 4 (4) | 2 (2) | 4 (4) | 2 (2) | 2 (3) | 1 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 3 (3) | 5 (5) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 12 (12) | 12 (12) | 10 (10) | 9 (9) | 2 (2) | 2 (2) | 12 (12) | 10 (10) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 6 (7) | 4 (4) | 4 (4) | 2 (2) | 2 (3) | 1 (2) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 4 (4) | 3 (3) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Leukopenia (Blood and lymphatic system disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Coagulopathy (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Haemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Monocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pancytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 2 (2) | 1 (1) | 0 (0)
Aortic valve incompetence (Cardiac disorders) | 2 (2) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Arrhythmia (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block (Cardiac disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiomegaly (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 3 (3) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
Supraventricular extrasystoles (Cardiac disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 4 (4) | 5 (5) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 1 (1) | 2 (2) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal infection (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1)
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug withdrawal syndrome neonatal (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperhidrosis (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 1 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oedema (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oedema peripheral (General disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Peripheral swelling (General disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Secretion discharge (General disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hypoalbuminaemia (Hepatobiliary disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bacteraemia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Klebsiella infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Base excess negative (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood lactate dehydrogenase increased (Investigations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood lactic acid increased (Investigations) | 1 (1) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0)
Blood pressure decreased (Investigations) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0)
Body temperature increased (Investigations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
C-reactive protein increased (Investigations) | 4 (4) | 5 (5) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 0 (0) | 3 (3) | 0 (0)
Cardiac output decreased (Investigations) | 3 (4) | 1 (1) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Coagulation time prolonged (Investigations) | 4 (4) | 1 (2) | 2 (2) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Fluid balance negative (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haematocrit decreased (Investigations) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 2 (2)
Hepatic enzyme decreased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oligurea (Renal and urinary disorders) | 6 (6) | 4 (4) | 3 (3) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 3 (3) | 1 (1)
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 4 (4) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Stridor (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4) | 3 (3) | 2 (2) | 3 (3) | 2 (2) | 2 (2) | 0 (0) | 2 (2) | 2 (2)

LIMITATIONS AND CAVEATS:
Data were significantly skewed due to differences in standard of care between US and non-US. The US dataset met the primary endpoint due to consistent early extubation in the OR. L-Citrulline promoted early extubation, reduced ventilator time & inotrope use in the US population. Post-hoc analyses gave a significant primary endpoint with an L-Citrulline therapeutic window of 100 µmol ±20% steady state concentration. A second Phase 3 RCT to be conducted in the US alone should confirm this result.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2017-08-11): https://cdn.clinicaltrials.gov/large-docs/37/NCT02891837/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/37/NCT02891837/SAP_001.pdf